CLINICAL TRIAL: NCT03461367
Title: Contemporary Chronic Total Occlusion Percutaneous Coronary Intervention Registry From Insight of Intravascular Ultrasound in Fuwai Hospital
Brief Title: CTO Registry From Insight of IVUS in Fuwai Hospital
Acronym: FWCTO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Lei Song, MD, Principal Investigator, China National Center for Cardiovascular Diseases
Other Study IDs: 20180223
Record Dates: First submitted 2018-03-03; First posted 2018-03-12 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Coronary Heart Disease; Chronic Total Occlusion of Coronary Artery; Percutaneous Coronary Intervention; Intravascular Ultrasound
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the long-term outcome of chronic total occlusion (CTO) patients underwent contemporary percutaneous coronary intervention (PCI) techniques, we design this single-center, large-sample, prospective registry with five-year clinical follow-up, based on the intravascular ultrasound (IVUS) finding.

DETAILED DESCRIPTION:
The study plan to include the patients with a CTO lesion in one of the three main epicardial coronary artery (diameter more than 2.5 mm) as the only target lesion. The CTO lesion is defined as 0 grade of thrombolysis in myocardial infarction (TIMI) flow with evidence of occlusion duration more than 3 months. All the PCI procedure will be performed by a group of certified operators in Fuwai Hospital, Beijing, China. All patients evaluate IVUS with automatic pullback (Opticross, Boston Scientific, US) performed after wire crossing. All the included patients are planned for five-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient >18 years old
* Thrombolysis in myocardial infarction trial (TIMI) 0 grade.
* Evidence of occlusion period more than 3 months.
* Patients eligible for PCI.
* Patients eligible for coronary artery bypass graft (CABG).
* Target vessel is one of the three main epicardial coronary arteries.

Exclusion Criteria:

* Acute myocardial infarction with ongoing ST-elevation
* Target vessel is left main or graft vessel.
* Target vessel diameter < 2.5 mm.
* Other situations ineligible for PCI judged in clinical practice.
* Left ventricular ejection fraction <30%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CTO Patients who underwent PCI with contemporary CTO techniques by certified operators in Fuwai Hospital.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Target vessel revascularization | 5-year follow-up after index PCI
  Any ischemic driven revascularization of the target vessel

SECONDARY OUTCOMES:
All-cause death | Within the first 1 month after PCI and during the 5-year follow-up
  Any cause of death
Cardiac death | Within the first 1 month after PCI and during the 5-year follow-up
  Cardiac death
Myocardial infarction | Within the first 1 month after PCI and during the 5-year follow-up
  Any myocardial infarction including perioperative MI
Stroke | Within the first 1 month after PCI and during the 5-year follow-up
  Ischemic or hemorrhagic stroke
Major adverse cardiac and cerebrovascular events (MACCE) | Within the first 1 month after PCI and during the 5-year follow-up
  Including all-cause death, myocardial infarction, stroke or any target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Bo Xu, Study Director — Fuwai Hospital, Catheter Lab
Locations (1):
- Lei Song, Beijing, Beijing Municipality, China